CLINICAL TRIAL: NCT02680262
Title: A Three-armed Randomised Controlled Trial of Non-participants in an Organised Cervical Cancer Screening Programme
Brief Title: Self-sampling for Non-participants in an Organised Cervical Cancer Screening Programme
Acronym: CHOiCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: af_randers
Record Dates: First submitted 2016-01-27; First posted 2016-02-11 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Cervical Cancer
Keywords: HPV self-sampling, cervical cancer screening
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intervention group 1 (Experimental): HPV self-sampling kit mailed directly
  Interventions: Behavioral: HPV self-sampling kit mailed directly
- Intervention group 2 (Experimental): HPV self-sampling kit on demand
  Interventions: Behavioral: HPV self-sampling kit on demand
- Intervention group 3 (Experimental): second reminder
  Interventions: Behavioral: Second reminder

INTERVENTIONS:
Behavioral: HPV self-sampling kit mailed directly — Women in intervention group 1 will be mailed a modified second reminder, a leaflet entitled Information about HPV self-sampling, and a self-sampling kit. The leaflet provides information about HPV and cervical cancer including benefits and harms about HPV self-sampling compared to regular screening. The kit includes a brush device (Evelyn Brush, Rovers Medical Devices B.V, Oss, Netherlands) to collect a cervico-vaginal sample for subsequent hrHPV testing, written and drawn instructions on how to obtain and mail the sample, and a pre-stamped return envelope addressed to the Department of Pathology, Randers Regional Hospital performing the hrHPV testing.
  Arms: Intervention group 1
Behavioral: HPV self-sampling kit on demand — Women in intervention group 2 receive the same material as arm 1, except for the kit, which will only be mailed to the women on demand. Additionally, the leaflet for this group contains information on how to order the kit.
  The modified second reminder in both intervention groups informs of the opportunity to collect a self-sample if wanted, but also about the opportunity to have a conventional specimen taken at a general practitioner (usual procedure).
  Arms: Intervention group 2
Behavioral: Second reminder — The standard second reminder informs women about the ongoing opportunity to have a conventional cervical sample taken by a general practitioner. (control group)
  Arms: Intervention group 3

SUMMARY:
The trial will evaluate the effect on participation in organised screening programme of a human papilloma virus (HPV) self-sampling kit directly mailed home or mailed on demand compared with the standard second reminder for regular screening.

DETAILED DESCRIPTION:
The CHOice trial is a parallel randomised controlled, open label trial. Participants will be equally randomised into three arms: 1) Directly mailed a second reminder including a HPV self-sampling kit; 2) Mailed a second reminder offering a HPV self-sampling kit, to be ordered by e-mail, by text message, by phone, or by website; and 3) Mailed a second reminder for a conventional practitioner-collected sample (control group).

ELIGIBILITY:
Inclusion Criteria:

* Women resident in the Central Denmark Region who have not participate in cervical cancer screening after an invitation and one reminder

Exclusion Criteria:

* Women younger than 30 years are not included due to the lower specificity of HPV DNA tests in younger women

Ages: 30 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9327 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Women who participate by returning a HPV self-sampling kit or having a practitioner-collected sample in the intervention groups compared to the proportion of women who have a practitioner-collected sample in the control group at 90 days after mail out. | 90 days
  Primary outcome will be the proportion of women who participate by returning a HPV self-sampling kit or having a practitioner-collected sample in the intervention groups compared to the proportion of women who have a practitioner-collected sample in the control group at 90 days after mail out.

SECONDARY OUTCOMES:
Women with a positive HPV self-collected sample who attend follow-up testing at 30, 60 or 90 days after mail out. | 30,60 or 90 days
  Secondary outcome will be the proportion of women with a positive HPV self-collected sample who attend follow-up testing at 30, 60 or 90 days after mail out of results

CONTACTS AND LOCATIONS:
Overall Officials: Mette Tranberg Nielsen, Phd Student, Principal Investigator — Department of Public Health Programmes
Locations (1):
- Mette Tranberg Nielsen, Randers, Randers NØ, Denmark

IPD SHARING:
Plan to Share IPD: No
The study is approved by the Danish Data Protection Agency, (j.no.:1-16-02-495-15)

REFERENCES:
- [Derived] Tranberg M, Bech BH, Blaakaer J, Jensen JS, Svanholm H, Andersen B. HPV self-sampling in cervical cancer screening: the effect of different invitation strategies in various socioeconomic groups - a randomized controlled trial. Clin Epidemiol. 2018 Aug 23;10:1027-1036. doi: 10.2147/CLEP.S164826. eCollection 2018. PMID 30197540
- [Derived] Tranberg M, Bech BH, Blaakaer J, Jensen JS, Svanholm H, Andersen B. Preventing cervical cancer using HPV self-sampling: direct mailing of test-kits increases screening participation more than timely opt-in procedures - a randomized controlled trial. BMC Cancer. 2018 Mar 9;18(1):273. doi: 10.1186/s12885-018-4165-4. PMID 29523108
- [Derived] Tranberg M, Bech BH, Blaakaer J, Jensen JS, Svanholm H, Andersen B. Study protocol of the CHOiCE trial: a three-armed, randomized, controlled trial of home-based HPV self-sampling for non-participants in an organized cervical cancer screening program. BMC Cancer. 2016 Nov 3;16(1):835. doi: 10.1186/s12885-016-2859-z. PMID 27809810